CLINICAL TRIAL: NCT02166242
Title: Phase 1c Single Arm Study of Thioredoxin Reductase Inhibitor Ethaselen, for the Treatment of Thioredoxin Reductase High Expressed Advanced Non-small Cell Lung Cancers Who Have Received More Than Two Lines Standard Treatment.
Brief Title: Ethaselen for the Treatment of Thioredoxin Reductase High Expression Advanced Non-small Cell Lung Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director of department of medical oncology, lung cancer and gastrointestinal cancer unit, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBSKE001
Record Dates: First submitted 2014-06-01; First posted 2014-06-18 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Carcinoma, Non-small Cell Lung
Keywords: non-small cell lung cancer; thioredoxin reductase
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — (1,2-bis(1,2-benzisoselenazolone-3(2H)-ketone))ethane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental (Experimental): patients pathologic diagnosis advanced non-small cell lung cancer who had received more than two lines standard treatment, according to NCCN Non-small cell lung cancer guideline, there were no standard treatment scheme for these patients. Approximately 40 patients will be included in the study, patients will received oral ethaselen dispersible tablet, 600 mg bid dose, patients may quit the study whenever they would like or investigator evaluate that progression disease has developed, or any grade of SAE developed during the study.
  Interventions: Drug: ethaselen

INTERVENTIONS:
Drug: ethaselen — ethaselen is a specific thioredoxin reductase inhibitor, which has finished phase 1a study in China, phase 1 study of ethaselen showed that 600 mg ethaselen bid could be well tolerated
  Other Names: BBSKE

SUMMARY:
Thioredoxin reductase plays an critical role in lung cancer patients, in vitro study showed that, ethaselen, specific inhibitor of thioredoxin reductase, could inhibit lung cancer cell growth and induce apoptosis. In China, phase 1 clinical trials of ethaselen showed that 1200 mg dose ethaselen could be well tolerated, in pre-clinical study we found that, approximately 50% non-small cell lung cancers harbored high thioredoxin reductase expression(IHC result ++ or +++), phase 1a/b of ethaselen had finished in 2008, the result showed that 1200mg ethaselen per day was safety and tolerated by Chinese malignant tumor patients.In pre-clinical research, our group found that, elevated of thioredoxin reductase activity was associated with the expression of thioredoxin reductase tested by immunohistochemistry, which means high expression of this enzyme may be a favourite predicted factor of ethaselen, the specific inhibitor of thioredoxin reductase.

DETAILED DESCRIPTION:
This phase 1c study will include patients pathologic diagnosis advanced non-small cell lung cancer who had received more than two lines standard treatment, according to NCCN Non-small cell lung cancer guideline, there were no standard treatment scheme for these patients. Approximately 40 patients will be included in the study, patients will received oral ethaselen dispersible tablet, 600 mg bid dose, primary endpoint of this study is 6 week disease control rate(DCR, CR+PR+SD), secondary endpoints include progression free survival(PFS), overall survival(OS), quality of life(QOL) and drug safety.

ELIGIBILITY:
Inclusion Criteria:

* advanced non-small cell lung cancer, stage IIIB/IV who had received more than 2 standard treatment scheme
* 18-75 years old, anticipate overall survival more than 3 months, ECOG 0-2
* within 4 weeks, not receive chemotherapy, radiotherapy or surgery
* HB≥90g/L； ANC ≥1.5×109/L；PLT ≥80×109/L
* EGFR/ALK mutation negative
* immunohistochemistry test of cancer tissue showed ++ or +++ of thioredoxin reductase
* brain metastasis without symptoms

Exclusion Criteria:

* according to NCCN non-small cell lung cancer guidelines (2014 v3), there were standard treatment scheme for the patients
* pregnancy or breast-feeding women
* any serious disease which could not be controled
* urine protein≥++, or 24h urine protein>1g
* received any anti-cancer treatment within 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
6 week disease control rate | within 6 weeks after patients received ethaselen treatment
  disease control rate will be measured within 6 weeks after patients received ethaselen treatment

SECONDARY OUTCOMES:
progression free survival | the first time investigator evaluate PFS will be at the sixth week since the study begin, the second time investigator evaluate PFS will be at the 12th week, the next time will be at the 18th week.
  the first time investigator evaluate PFS will be at the sixth week since the study begin, the second time investigator evaluate PFS will be at the 12th week, the next time will be at the 18th week. Up to 30 weeks after the study was finished.
overall survival | the first time investigator evaluate OS will be at the sixth week since the study begin, the second time investigator evaluate PFS will be at the 12th week, the next time will be at the 18th week. Up to 30 weeks after the study was finished.
  the first time investigator evaluate OS will be at the sixth week since the study begin, the second time investigator evaluate OS will be at the 12th week, the next time will be at the 18th week. Up to 30 weeks after the study was finished.
safety of drug | safety of drug will be recorded during treatment, up to 6 weeks after treatment
  any SAE should be recorded and reported to SFDA within 1 day during ethaselen treatment, after treatment drug associated safety will be in 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, MD, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- Hunan province tumor hospital, Changsha, Hunan, China

REFERENCES:
- [Background] Wang L, Yang Z, Fu J, Yin H, Xiong K, Tan Q, Jin H, Li J, Wang T, Tang W, Yin J, Cai G, Liu M, Kehr S, Becker K, Zeng H. Ethaselen: a potent mammalian thioredoxin reductase 1 inhibitor and novel organoselenium anticancer agent. Free Radic Biol Med. 2012 Mar 1;52(5):898-908. doi: 10.1016/j.freeradbiomed.2011.11.034. Epub 2011 Dec 21. PMID 22210352
- [Background] Wang L, Fu JN, Wang JY, Jin CJ, Ren XY, Tan Q, Li J, Yin HW, Xiong K, Wang TY, Liu XM, Zeng HH. Selenium-containing thioredoxin reductase inhibitor ethaselen sensitizes non-small cell lung cancer to radiotherapy. Anticancer Drugs. 2011 Sep;22(8):732-40. doi: 10.1097/CAD.0b013e32834618bc. PMID 21562407
- [Background] Poerschke RL, Moos PJ. Thioredoxin reductase 1 knockdown enhances selenazolidine cytotoxicity in human lung cancer cells via mitochondrial dysfunction. Biochem Pharmacol. 2011 Jan 15;81(2):211-21. doi: 10.1016/j.bcp.2010.09.024. Epub 2010 Oct 12. PMID 20920480
- [Background] Zhao F, Yan J, Deng S, Lan L, He F, Kuang B, Zeng H. A thioredoxin reductase inhibitor induces growth inhibition and apoptosis in five cultured human carcinoma cell lines. Cancer Lett. 2006 May 8;236(1):46-53. doi: 10.1016/j.canlet.2005.05.010. Epub 2005 Jun 27. PMID 15982805
- [Background] Fu JN, Li J, Tan Q, Yin HW, Xiong K, Wang TY, Ren XY, Zeng HH. Thioredoxin reductase inhibitor ethaselen increases the drug sensitivity of the colon cancer cell line LoVo towards cisplatin via regulation of G1 phase and reversal of G2/M phase arrest. Invest New Drugs. 2011 Aug;29(4):627-36. doi: 10.1007/s10637-010-9401-y. Epub 2010 Mar 2. PMID 20195699
- [Background] Tan Q, Li J, Yin HW, Wang LH, Tang WC, Zhao F, Liu XM, Zeng HH. Augmented antitumor effects of combination therapy of cisplatin with ethaselen as a novel thioredoxin reductase inhibitor on human A549 cell in vivo. Invest New Drugs. 2010 Jun;28(3):205-15. doi: 10.1007/s10637-009-9235-7. Epub 2009 Mar 7. PMID 19271154